CLINICAL TRIAL: NCT03947723
Title: Histologic Evaluation Comparing Power Settings in Radiofrequency Ablation on Eyelash Follicles
Brief Title: Histology Evaluation of Radiofrequency Ablation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Left Institution
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: STUDY00000551; LSU IRB (Other: 19-016)
Record Dates: First submitted 2019-05-07; First posted 2019-05-13 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Trichiasis
Keywords: trichiasis; radiofrequency ablation; epilation; histology
MeSH Terms: conditions — Trichiasis | interventions — Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: This will be a modified factorial trial. The tissue from all patients will be divided into 4 sections and undergo radiofrequency ablation at different settings in each section, giving us 4 groups. These 4 groups will be compared to each other.
Who Masked: Outcomes Assessor
Masking Description: The person examining the slides will be blinded to the power setting used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Low power (Experimental): These tissue sections will receive radiofrequency ablation to each eyelash follicle at a power of "low."
  Interventions: Device: Radiofrequency ablation
- 1 power (Experimental): These tissue sections will receive radiofrequency ablation to each eyelash follicle at a power of 1.
  Interventions: Device: Radiofrequency ablation
- 1.5 power (Experimental): These tissue sections will receive radiofrequency ablation to each eyelash follicle at a power of 1.5
  Interventions: Device: Radiofrequency ablation
- 2 power (Experimental): These tissue sections will receive radiofrequency ablation to each eyelash follicle at a power of 2.
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Device: Radiofrequency ablation — The eyelid segments to be excised as part of their planned lateral tarsal strip procedure will be marked and divided into 4 equal sections (2 sections on each lid). A corneal shield will be placed into the fornix prior to treatment. Each section will be treated with the designated power setting in the following manner. The probe will be inserted into the follicle under direct visualization to a depth of approximately 1.4 mm. The designated power will be applied for 1 second. All lashes in each segment will be treated. The segments will then be excised and placed into labelled and coded containers of formalin.

SUMMARY:
Trichiasis is a disorder of misdirected eyelashes in which the lashes grow inward towards the eye. Trichiasis can occur as a result of chronic inflammation, infection, such as in herpes or trachoma, trauma, or rare diseases like ocular cicatricial pemphigoid or Stevens-Johnson syndrome. Trichiasis can result significant pain and corneal compromise, ranging from punctate erosions to frank abrasions, as the lashes constantly contact and irritate the ocular surface. Several treatment modalities are available, including mechanical epilation, electroepilation, cryotherapy, laser therapy, and surgical procedures to redirect the lashes. Radiofrequency ablation is a type of electroepilation that utilizes radiowaves to heat and destroy hair follicles. A fine needle is inserted into the follicle and current is applied to destroy the follicle. The needle allows the energy to be focused into the follicle and limits scarring of the surrounding tissues, and the follicles are in theory permanently destroyed in this procedure. Success rates are variable however, ranging from 56 to 90%. Currently, there is no standardized protocol for performing radiofrequency ablation. Many practitioners choose their power settings based on experience, and the Ellman Surgitron machine, a commonly used radiofrequency unit, actually states in their instructions that the power should be titrated based on user experience. In the literature, settings anywhere from 1 to 3 are seen. In this study, our purpose is to examine the effects of different power settings in radiofrequency at the histologic level. The investigators plan to test different power settings on eyelid tissue that would be normally excised and discarded during eyelid correction surgeries. The investigators hope to determine if there is an ideal power setting to achieve hair follicle destruction while minimizing surrounding tissue damage, which could then be used as the standard power setting for radiofrequency ablation of trichiatic lashes in clinical practice. The investigators hypothesize that as power increases, the extent and severity of tissue damage will increase.

DETAILED DESCRIPTION:
Subject fulfilling the inclusion and exclusion criteria and willing to participate in the study will be enrolled. All participants will receive all 4 treatments at the varying power settings (low, 1, 1.5, 2).

The patients will be prepped for their surgery in the usual fashion. This portion of the procedure is not experimental and is an elective surgery that the patients are choosing to undergo prior to enrolling in the study. This procedure is performed in the operating room. After adequate anesthesia is achieved, subcutaneous 2% lidocaine with epinephrine with 0.5% marcaine, and vitrase is injected into the lower eyelids and lateral canthal areas. The face is prepped and draped in sterile fashion using topical Betadine. A corneal shield will be placed into the fornix at this time. A lateral canthal incision is then made using a #15 blade. Straight Stevens scissors are used to perform a canthotomy and monopolar cautery was used to incise the inferior crus of the lateral canthal tendon. Hemostasis is maintained. The freed lower eyelid is draped over the zygoma. The excess eyelid is then excised full-thickness with Westcott scissors. (If this excess eyelid skin is at least 5 mm on both sides, the study will be performed and the treatments will be applied at this point). The tissue will be marked and divided into 4 equal sections (2 sections on each lid). Each section will be treated with the designated power setting in the following manner.

The probe will be inserted into the follicle under direct visualization to a depth of approximately 1.4 mm. The designated power will be applied for 1 second. All lashes in each segment will be treated. The segments will then be excised and placed into labelled and coded containers of formalin.

Attention will then be directed back to completing the lateral tarsal strip/eyelid surgery. The remainder of the surgery will be performed in the usual fashion and is not part of the experimental portion of the study. One 4-0 Vicryl on P-2 needle is then passed through the tarsus backhanded anterior inferiorly exiting posterior superiorly within the wound and then passed back through the periosteum approximately 3 mm from the orbital rim at the level of the superior crus of the lateral canthal tendon and temporarily tied. This procedure is repeated in full on the other side. The sides are compared. Once the proper contour and tightness is achieved, the suture is permanently tied in a horizontal mattress fashion after passing back through the remnants of the inferior crus. Attention is then turned to the upper lid, whose lateral mucocutaneous junction is trimmed using Westcott scissors. The gray lines of the lateral upper and lower eyelids arre reapposed using 6-0 Vicryl. The lateral canthal incisions are closed with a running 6-0 Prolene suture. Tobradex ointment is applied to the eye and eyelid. The patient is awakened and extubated and taken to the recovery room in stable condition. The patients will be examined at their post-operative week 1 and month 1 visits as per the usual standard of care. After the 1 month visit, their participation in the study is complete.

The tissue sections will be sent to the pathology department for sectioning and staining. The tissue will be sectioned through the follicles. The slides will be stained with hemotoxylin and eosin and Masson-Trichrome. The extent of tissue damage will be measured as the diameter of abnormal/damaged tissue in microns. The severity will be graded on a numerical scale from 0-3. The results will be compared among the 4 power settings.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing the bilateral tarsal strip procedure
* The procedure requires at least 5 mm of tissue to be excised from each side to provide adequate tightening of the lower eyelids (to be determined intra-operatively)
* Caucasian (to control for any different responses ellicited by the treatment in pigmented skin)

Exclusion Criteria:

* previous treatments for trichiasis along the lateral lower eyelid
* madarosis of eyelashes
* hypertrichosis of eyelashes
* patients undergoing only unilateral tarsal strip procedures
* history of eyelid trauma or chemical burns
* patients with a history of disorders affecting the mucus membranes (ie: Stevens-Johnson syndrome, ocular cicatricial pemphigoid)
* history of eyelid surgery
* history of facial skin cancers
* patients with eyelid lesions affecting the lateral lower eyelids
* patients with active inflammatory ocular diseases (keratitis, scleritis, conjunctivitis, etc).

These exclusion criteria are to generally encompass and exclude any eyelid or eyelash pathology that may confuse what histology changes are from the study treatments versus what pathology was already there at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Extent of tissue damage | Through study completion, approximately 6 months
  The extent of damage will be measured on the tissue sections. The diameter of abnormal/damaged tissue will be measured in microns.
Severity of tissue damage | Through study completion, approximately 6 months
  The severity will be graded on a scale from 0 to 3, with 0 being no tissue changes and going up to 3 which will represent severe tissue changes.

CONTACTS AND LOCATIONS:
Overall Officials: Priya Sahu, MD, Principal Investigator — Ochsner Health System; Jayne Weiss, MD, Principal Investigator — Louisiana State University Health Sciences Center

IPD SHARING:
Plan to Share IPD: No
No plan to share with other researchers

REFERENCES:
- [Background] Nakamoto, D., Bernardino, C.R. The Annoying Lash in the Eye: A Review of Trichiasis. Review of Ophthalmology. Retrieved from: https://www.reviewofophthalmology.com/article/the-annoying-lash-in-the-eye-a-review-of-trichiasis. 2007.
- [Background] Kim GN, Yoo WS, Kim SJ, Han YS, Chung IY, Park JM, Yoo JM, Seo SW. The effect of 0.02% mitomycin C injection into the hair follicle with radiofrequency ablation in trichiasis patients. Korean J Ophthalmol. 2014 Feb;28(1):12-8. doi: 10.3341/kjo.2014.28.1.12. Epub 2014 Jan 21. PMID 24505196
- [Background] Kezirian GM. Treatment of localized trichiasis with radiosurgery. Ophthalmic Plast Reconstr Surg. 1993 Dec;9(4):260-6. doi: 10.1097/00002341-199312000-00006. PMID 8305373